CLINICAL TRIAL: NCT07015034
Title: Developing and Testing a Model to Identify Preventive Vision Loss Among Older Patients in General Practice (DETECT)
Brief Title: Developing and Testing a Model to Identify Preventive Vision Loss Among Older Patients in General Practice
Acronym: DETECT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Catharina Thiel Sandholdt, Assistant Professor, University of Copenhagen
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: 869353; 869353 (Other Grant/Funding Number: Velux Foundation)
Record Dates: First submitted 2025-05-20; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Vision Impairment and Blindness; Glaucoma; Age-Related Macular Degeneration; Cataract; Diabetic Retinopathy
MeSH Terms: conditions — Vision Disorders; Blindness; Glaucoma; Macular Degeneration; Cataract; Diabetic Retinopathy

STUDY DESIGN:
Masking Description: GP's or GP nurses, optometrists and the project ophtalmologist all give their anamnesis (and potential diagnosis). Their anamnesis are blinded to each other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Three vision tests in general practice (Other): All patients recruited in general practice are asked to fill out a patient questionnaire and examined:
  - Collenbrander Mixed contrast card: testing near vision binocularly at 40 cm, using both 100% and 10% contrast.
  - Amsler Test: Conducted for both eyes to check for central vision issues.
  - Visual Field Test: Performed using the Donders method to assess peripheral vision, conducted for both eyes.
  After tests in general practice, all patients undergo a comprehensive vision assessment at local optician shops, which include the following tests:
  * Habitual Vision Testing: Near and distance vision with habitual glasses.
  * Best Corrected Distance Vision: Monocular and binocular.
  * Intraocular Pressure Measurement Assessed using air tonometry or Icare.
  * Ocular Imaging: 3D peripapillary and macula optical coherence tomography (OCT) scans, and fundus photography.
  A project ophtalmologist analyze patient-data from optometrists.
  Interventions: Other: focus on vision impairment in older patients in general practice

INTERVENTIONS:
Other: focus on vision impairment in older patients in general practice — GP or GP nurse carry out the three vision tests. All patients visit optician shop collaborating with the project. An ophthalmologist review data from optometrists and provide an epicrisis to general practice. In case of acute conditions, the ophthalmologist is responsible for expedient treatment. If the patient needs further control by ophthalmologist within 12 month waiting time, general practice are responsible for referring the patient.

SUMMARY:
In this cohort study, the investigators will test vision screenings in Danish general practice for patients over 70 years of age with minimum one chronic condition. The main outcome is detection of vision impairment and secondary outcome is detection of conditions needing ophthalmologic follow-up but not presenting vision impairment at present time.

DETAILED DESCRIPTION:
Introduction: The number of people living with visual impairment is increasing. Visual impairment causes loss in quality of life and reduce self-care abilities. The burden of disease is heavy for people experiencing visual impairment and their relatives. The severity and progression of age-related eye diseases are dependent on the time of detection and treatment options, making timely access to healthcare critical in reducing visual impairment. General practice plays a key role in public health by managing preventive healthcare, diagnostics and treatment of chronic conditions. General practitioners (GPs) coordinate services from other healthcare professionals. More involvement of the primary sector could potentially be valuable in detecting visual impairment.

Methods: Investigators apply the Medical Research Council framework for complex interventions to develop a primary care intervention with the GP as a key actor, aimed at identifying and coordinating care for patients with low vision. The development process will engage patients, relatives and relevant health professional stakeholders. The investigators will pilot test the feasibility of the intervention in a real-world general practice setting. The intervention model will be developed through a participatory approach using qualitative and creative methods such as graphical facilitation. The project aims to explore the potentials and limitations of general practice in relation to detection of preventable vision loss.

Ethics and dissemination: Ethics approval is obtained from local authority and the study meets the requirements from the Declaration of Helsinki. Dissemination is undertaken through research papers and to the broader public through podcasts and patient organisations.

ELIGIBILITY:
Inclusion Criteria:

* +70 years
* One or more chronic diseases
* Are followed by GP du to chronic disease

Exclusion Criteria:

* Dementia diagnosis
* Known eye-diseases or are currently followed by private ophtalmologist
* Not able to understand Danish

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 460 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2027-07-15 (Estimated)

PRIMARY OUTCOMES:
vision below 0,7 habitual vision on the best seeing eye | From enrollment in GP setting and diagnostic tests to ophtalmologist review two weeks hereafter
  The main outcome is detected vision impairment defined as a vision below 0,7 habitual vision on the best seeing eye with both eyes open wearing their current glasses if any

SECONDARY OUTCOMES:
detection of eye-diseases | From enrollment in GP setting and diagnostic tests to ophtalmologist review two weeks hereafter
  Secondary outcome is detected eye-diseases and changes in the eye or retina causing a potential vision impairment on a later stage. Investigators specifically screen for glaucoma, cataract, age-related macular degeneration (AMD), but other conditions can be detected as well.

CONTACTS AND LOCATIONS:
Overall Officials: Frans B Waldorff, Principal Investigator — Center for Almen Medicin, KU
Locations (2):
- Denmark (2):
  - Søndre Lægehus (GP practice), Køge, Køge
  - Louise Uhre General Practice, Køge

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sandholdt CT, Jonsson ABR, Reventlow S, Bach-Holm D, Line K, Kolko M, Jacobsen MH, Mathiesen OH, Waldorff FB. DETECT: DEveloping and testing a model to identify preventive vision loss among older paTients in gEneral praCTice - protocol for a complex intervention in Denmark. BMJ Open. 2023 May 29;13(5):e069974. doi: 10.1136/bmjopen-2022-069974. PMID 37247966